CLINICAL TRIAL: NCT00327171
Title: A Multicenter, Randomized, Double-blind, Parallel-arm, Two-stage Study of the Efficacy and Safety of AVE0005 (VEGF Trap) Administered Intravenously Every 2 Weeks in Patients With Platinum-resistant and topotecan-and/or Liposomal Doxorubicin-resistant Advanced Ovarian Cancer
Brief Title: Study of AVE0005 (VEGF Trap) in Patients With Chemoresistant Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARD6122; AVE0005
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Neoplasms; Cancer of the Ovary
Keywords: ovarian cancer; angiogenesis; angiogenesis inhibition; VEGF-Trap fusion recombinant protein; Cancer and other neoplasms
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept 2.0 mg/kg (Experimental): Participants with advanced ovarian epithelial adenocarcinoma administered 2.0 mg/kg Aflibercept.
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)
- Aflibercept 4.0 mg/kg (Experimental): Participants with advanced ovarian epithelial adenocarcinoma administered 4.0 mg/kg Aflibercept.
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)

INTERVENTIONS:
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — Aflibercept 4.0 mg/kg administered intravenously (IV) over 1 hour once every 2 weeks.
  Aflibercept could be reduced by 1 dose level ( to 2.0 mg/kg) or 2 dose levels (to 1.0 mg/kg) in case of uncontrolled hypertension or urinary protein >3.5 g/24 hours. Intrapatient dose escalation was not to be permitted. Participants requiring more than 2 dose level reductions would be withdrawn from study treatment.
  Arms: Aflibercept 4.0 mg/kg
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — Aflibercept 2.0 mg/kg administered intravenously (IV) over 1 hour once every 2 weeks.
  Aflibercept could be reduced by 1 dose level (to 1.0 mg/kg) or 2 dose levels (to 0.5 mg/kg) in case of uncontrolled hypertension or urinary protein >3.5 g/24 hours. Intrapatient dose escalation was not to be permitted. Participants requiring more than 2 dose level reductions would be withdrawn from study treatment.
  Arms: Aflibercept 2.0 mg/kg

SUMMARY:
This study evaluated outcomes in participants with advanced ovarian epithelial adenocarcinoma receiving aflibercept.

The primary objective was to compare the objective response rate of Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) 4.0 mg/kg and 2.0 mg/kg, administered intravenously (IV) every 2 weeks with historical control in participants with advanced ovarian epithelial (including fallopian tube and primary peritoneal) adenocarcinoma resistant to platinum and topotecan and/or liposomal doxorubicin.

The secondary objectives was to further assess efficacy, safety, pharmacokinetics, potential biological and pharmacogenomic markers of study drug activity, and health-related quality of life.

This study employed an Independent Review Committee (IRC) for radiological tumor assessments. For all tumor assessment-related efficacy variables, two analyses were performed: the primary analysis was based on Independent Review Committee (IRC) reviewed data and the secondary analysis was based on Investigator evaluation. If an endpoint was evaluated by the IRC, the IRC reviewed data is reported for this study.

DETAILED DESCRIPTION:
The study included:

* A screening period for 21 days
* Randomization at baseline (Treatment was initiated with 5 days of randomization)
* A treatment period with 14-day study treatment cycles until a study withdrawal criterion was met
* A follow-up period up to 60 days after the end of treatment

Withdrawal criteria that led to treatment discontinuation were:

* The participant or their legally authorized representative requested to withdraw
* In the investigator's opinion, continuation of the study would be detrimental to the participant's well being, due to reasons such as disease progression, unacceptable toxicity, noncompliance, or logistical considerations.
* A specific request by the Sponsor
* Participant had intercurrent illness that prevented further administration of study treatment
* Participant had more than 2 aflibercept dose reductions
* Participant had arterial thromboembolic events, including cerebrovascular accidents, myocardial infarctions, transient ischemic attacks, new onset or worsening of pre-existing angina
* Participant had radiographic evidence of intestinal obstruction (e.g., dilated loops of bowel accompanied by air-fluid levels) or gastrointestinal perforation (e.g., presence of extraluminal gas) requiring surgical intervention
* Participant was lost to follow-up

After discontinuing treatment, participants remained on the study until the last post-treatment visit or until recovery of drug related toxicities, whichever was later.

ELIGIBILITY:
Participants who met the following criteria were eligible for the study.

Inclusion Criteria:

* Histologically-confirmed ovarian epithelial (including fallopian tube and primary peritoneal) adenocarcinoma.
* Prior treatment with at least 2 treatment regimens in the advanced disease treatment setting
* Platinum-resistant disease defined by relapse or progression of disease during or after treatment, or drug intolerance
* Topotecan- and/or liposomal doxorubicin-resistant disease defined by relapse or progression of disease during or after treatment, or drug intolerance
* Evidence of at least one unidimensional measurable tumor lesion by computed tomography (CT) or magnetic resonance imaging (MRI) scan according to Response Evaluation Criteria in Solid Tumors (RECIST) that has not been treated with surgery or radiation therapy

Exclusion Criteria:

* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or for in situ carcinoma of the cervix uteri
* Prior treatment with a vascular endothelial growth factor (VEGF) or VEGF receptor inhibitor
* More than 3 chemotherapy regimens in the advanced disease treatment setting
* Uncontrolled hypertension

The above information is not intended to contain all considerations relevant to potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland

REFERENCES:
- [Result] Tew WP, Colombo N, Ray-Coquard I, Del Campo JM, Oza A, Pereira D, Mammoliti S, Matei D, Scambia G, Tonkin K, Shun Z, Sternas L, Spriggs DR. Intravenous aflibercept in patients with platinum-resistant, advanced ovarian cancer: results of a randomized, double-blind, phase 2, parallel-arm study. Cancer. 2014 Feb 1;120(3):335-43. doi: 10.1002/cncr.28406. Epub 2013 Oct 11. PMID 24127346
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 218 participants were randomized in this study. Three participants in the 2 mg/kg treatment group did not receive any study medication.
Groups:
- Aflibercept 2.0 mg/kg: Participants with advanced ovarian epithelial adenocarcinoma administered 2.0 mg/kg Aflibercept intravenously every two weeks
- Aflibercept 4.0 mg/kg: Participants with advanced ovarian epithelial adenocarcinoma administered 4.0 mg/kg Aflibercept intravenously every two weeks
Period: Overall Study
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Started | 109 | 109
Completed | 1 (Participants received treatment until they met treatment discontinuation criteria) | 0 (Participants received treatment until they met treatment discontinuation criteria)
Not Completed | 108 | 109
Not completed — Did not receive study medication | 3 | 0
Not completed — Adverse Event | 23 | 23
Not completed — Disease progression/lack of efficacy | 68 | 69
Not completed — Investigator/participant request | 1 | 8
Not completed — Clinical progression | 12 | 8
Not completed — Undisclosed history of ischemia | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg | Total
Number analyzed (Participants) | 109 | 109 | 218
Age, Customized [Number; unit: participants]
  <35 years | 3 | 3 | 6
  >=35 to <45 years | 10 | 6 | 16
  >=45 to <55 years | 21 | 25 | 46
  >=55 to <65 years | 37 | 43 | 80
  >=65 to <75 years | 32 | 25 | 57
  >=75 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 109 | 218
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 104 | 107 | 211
  Black | 3 | 1 | 4
  Asian, Oriental | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Based on the Analysis by an Independent Review Committee (IRC) - Simon's Cohort
Description: OR included Complete Response (CR) and Partial Response (PR). Per RECIST, CR was disappearance of all target or non-target lesions, or normalization of tumor marker levels (for non-target lesions) and PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, with baseline sum LD as reference.
  Tumors were assessed by an independent third-party core imaging laboratory evaluating the chest, abdomen, and pelvis by Computerized Tomography (CT) scans or Magnetic Resonance Imaging (MRI) scans; and responses were confirmed by repeat tumor imaging 4-6 weeks later.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: Simon's cohort: The first 67 evaluable participants, based on Simon's two-stage design that required 67 evaluable participants per group to maintain a targeted 80% power for Objective response rate versus historical controls.
Measure: Number; unit: participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 67 | 67
participants | 0 | 3

2. Secondary Outcome: Number of Participants With a Clinical Benefit Response (CBR) as Per RECIST Based on the Analysis by the IRC
Description: CBR was defined as having a Stable disease (SD) for >= 6 months or a confirmed OR (PR or CR). Based on RECIST:
  * SD was neither a sufficient shrinkage of the target lesions to qualify for PR nor sufficient increase to qualify for Progressive disease (PD), the persistence of non-target lesions or the maintenance of tumor marker level above the normal limits (for non-target lesions)
  * CR was the disappearance of all target or non-target lesions; and PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, with reference to the baseline sum LD.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 67 | 67
participants | 12 | 7

3. Secondary Outcome: Duration of Response (DR) Based on the Analysis by an Independent Review Committee (IRC)
Description: DR was defined as the time interval from the first documentation of CR or PR to the date of tumor progression (or disease progression) as determined by RECIST, or death from any cause, whichever was earlier.
  Based on RECIST, progressive disease was at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, the appearance of one or more new target or non-target lesions, or the unequivocal progression of existing non-target lesions.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: Efficacy evaluable population: All participants with advanced ovarian epithelial carcinoma who were randomized, underwent baseline tumor assessment, and received at least part of one dose of aflibercept.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 1 | 5
days | 164 (NA) — NA: Not calculable since only one participant achieved CR or PR | 149.8 (70.4)

4. Secondary Outcome: Tumor Marker Response Rate (TMRR) Based on the Gynecologic Cancer Intergroup (GCIG) Definition
Description: TMRR was the proportion of evaluable participants achieving a cancer antigen -125 (CA-125) response based on GCIG definition. A response to CA-125 occurred if after two elevated levels before therapy there was at least a 50% decrease in a post-treatment serum sample, which was confirmed by an independent sample collected 21 days or later that was =< 110% of the post-treatment serum sample.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: Randomized participants who received at least part of one dose of aflibercept, had a baseline tumor assessment, had a valid CA-125 assessment (requiring at least two pretreatment sample and 2 post-treatment samples), did not receive mouse antibodies and had no medical or surgical interference with their peritoneum or pleura in the previous 28 days.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 61 | 69
percentage of participants | 11.5 [4.7 to 22.2] | 11.6 [5.1 to 21.6]

5. Secondary Outcome: Time to Tumor Progression (TTP) as Per RECIST Based on the Analysis by the IRC
Description: TTP was defined as the time interval measured from the date of randomization to the date of tumor progression as determined by RECIST. TTP was estimated from Kaplan-Meier curves.
  For a participant who did not reach tumor progression during study, the censoring date was the date of the last valid tumor burden assessment or the date of study cut-off, whichever was earlier. If the participant had no valid post-baseline tumor burden assessment due to early termination, the censoring date was the date of randomization.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: Tumor Progression Events
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
Number analyzed (Tumor Progression Events) | 66 | 66
weeks | 13.1 [12.1 to 16.7] | 12.7 [12 to 18.9]
Statistical Analysis 1: Comparison: Aflibercept 2.0 mg/kg vs Aflibercept 4.0 mg/kg; Test type: Superiority or Other; p = 0.5043, Log Rank; Hazard Ratio (HR) = 1.123, 95% CI 2-sided [0.80 to 1.58] — Estimated using Cox proportional Hazard model using treatment as the factor

6. Secondary Outcome: Time to Tumor Marker (CA-125) Progression (TTMP)
Description: TTMP was the time interval from the date of randomization to the date of tumor marker progression as was defined by GCIG for the evaluable participants. TTMP was estimated using Kaplan-Meier curves.
  For a participant who did not reach tumor marker progression (TMP) during study, the censoring date was the date of the last valid tumor burden assessment or the date of study cut-off, whichever was earlier. If the participant had no valid post-baseline tumor burden assessment due to early termination, the censoring date was the date of randomization.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: Participants with a valid assessment of CA-125 (requiring at least one pretreatment sample and 2 post-treatment samples).
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: Tumor Marker Progression events
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 76 | 84
Number analyzed (Tumor Marker Progression events) | 15 | 20
weeks | NA [24.1 to NA] — The value was not calculable due to the limited number of events. | NA [22.7 to NA] — The value was not calculable due to the limited number of events.

7. Secondary Outcome: Number of Participants With Disease Progression Events for Progression-free Survival (PFS) Analysis by the IRC.
Description: PFS was as the time interval measured from the date of randomization to the date of tumor progression as determined by RECIST or death from any cause, whichever was earlier.
  The number of participants with tumor/disease progression are reported. Participants who did not reach tumor progression during study, or had no valid post-baseline tumor burden assessment due to early termination, were censored in the PFS analysis.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
participants
  With disease progression as the first event | 66 | 66
  Death without disease progression | 16 | 23
  Censored due to drop-out | 18 | 14
  Censored at study cut-off | 6 | 6

8. Secondary Outcome: Progression-free Survival (PFS) Time Based on Analysis by the IRC
Description: PFS was as the time interval measured from the date of randomization to the date of tumor progression as determined by RECIST or death from any cause, whichever was earlier. PFS was estimated using Kaplan-Meier curves.
  For a participant who did not reach tumor progression during study, the censoring date was the date of the last valid tumor burden assessment or the date of study cut-off, whichever was earlier. If the participant had no valid post-baseline tumor burden assessment due to early termination, the censoring date was the date of randomization.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: PFS Events
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
Number analyzed (PFS Events) | 82 | 89
weeks | 13.0 [11.7 to 16.7] | 13.3 [11.2 to 18.9]
Statistical Analysis 1: Comparison: Aflibercept 2.0 mg/kg vs Aflibercept 4.0 mg/kg; Test type: Superiority or Other; p = 0.5592, Log Rank; Hazard Ratio (HR) = 1.093, 95% CI 2-sided [0.81 to 1.48] — Estimated using Cox proportional Hazard model using treatment as the factor (4mg/kg vs. 2mg/kg)

9. Secondary Outcome: Overall Survival (OS) Time
Description: OS was the time interval between randomization and the date of death from any cause. OS was estimated using Kaplan-Meier curves
  A participant was censored for the OS analysis if the participant were alive during the study. The censoring date was either at the date that the participant was last known to be alive or the date of study cut-off, whichever was earlier.
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: Events (Death)
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
Number analyzed (Events (Death)) | 50 | 58
weeks | 59.0 [41.6 to 84.1] | 49.3 [37.4 to 62.7]
Statistical Analysis 1: Comparison: Aflibercept 2.0 mg/kg vs Aflibercept 4.0 mg/kg; Test type: Superiority or Other; p = 0.5457, Log Rank; Hazard Ratio (HR) = 1.124, 95% CI 2-sided [0.77 to 1.64] — Estimated using Cox proportional Hazard model using treatment as the factor (4 mg/kg vs. 2mg/kg)

10. Primary Outcome: Number of Participants With Confirmed Objective Response (OR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Based on the Analysis by the IRC - Efficacy Evaluable Population
Description: as for outcome 1
Time Frame: From enrollment to efficacy cut-off date, 18 January 2008 (approximately 20 months)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
participants | 1 | 5

11. Secondary Outcome: Overall Safety - Number of Participants With Adverse Events (AE)
Description: All AEs regardless of seriousness or relationship to study treatment, spanning from the first administration of study treatment until 30 days after the last administration of study treatment, were recorded, and followed until resolution or stabilization. The number of participants with all treatment emergent adverse events (TEAE), serious adverse events (SAE), TEAE leading to death, and TEAE leading to permanent treatment discontinuation are reported.
Time Frame: up to 30+/-5 days after treatment discontinuation, or up to recovery or stabilization of a followed-up adverse event
Population: Safety population: All randomized participants who received at least part of one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 106 | 109
participants
  With any TEAE | 106 | 108
  With any serious TEAE | 50 | 55
  With any TEAE leading to death | 14 | 14
  With TEAE leading to treatment discontinuation | 23 | 24

12. Secondary Outcome: Participant's Assessment of Health Related Quality of Life (HRQL) Using a by Using the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) Questionnaire
Description: The FACT-O questionnaire consists of 38 scored questions (scored from 0-4) that address physical well-being, social/family well-being, emotional well-being, functional well-being and some additional concerns which relate specifically to ovarian cancer symptoms. For each question, higher scores reflect a better quality of life. The total FACT-O score ranges from 0-152, with 152 indicating the best outcome.
Time Frame: On Day 1 of Cycle 1 (baseline) , and after Day 14 of Cycle 2
Population: All randomized participants who had evaluable FACT-O questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 97 | 104
score on a scale
  Baseline (N=97, N=104) | 105.3 (20.0) | 101.1 (22)
  Change (baseline to Cycle 2-Day 14) (N=79, N=77) | -1.1 (12.7) | -2.8 (13.9)

ADVERSE EVENTS:
Time Frame: From treatment initiation to June 9, 2010
Description: Safety population: All randomized participants who received at least part of one dose of study treatment.
Arm/Group | Aflibercept 2.0 mg/kg | Aflibercept 4.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 51/106 | 56/109
Other Adverse Events (participants affected / at risk) | 105/106 | 106/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept 2.0 mg/kg (N=106) | Aflibercept 4.0 mg/kg (N=109)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6
Ascites (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 10 | 6
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 2
Disease progression (General disorders) | 3 | 7
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 2
Sudden death (General disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Hepatitis a (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 3 | 3
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 6
Phlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept 2.0 mg/kg (N=106) | Aflibercept 4.0 mg/kg (N=109)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 36 | 40
Abdominal pain upper (Gastrointestinal disorders) | 14 | 17
Constipation (Gastrointestinal disorders) | 37 | 27
Diarrhoea (Gastrointestinal disorders) | 31 | 39
Dry mouth (Gastrointestinal disorders) | 6 | 4
Intestinal obstruction (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 44 | 43
Stomatitis (Gastrointestinal disorders) | 10 | 8
Toothache (Gastrointestinal disorders) | 9 | 7
Vomiting (Gastrointestinal disorders) | 38 | 30
Asthenia (General disorders) | 30 | 27
Fatigue (General disorders) | 42 | 44
Mucosal inflammation (General disorders) | 13 | 19
Oedema peripheral (General disorders) | 12 | 12
Pyrexia (General disorders) | 18 | 21
Nasopharyngitis (Infections and infestations) | 7 | 9
Urinary tract infection (Infections and infestations) | 13 | 5
Weight decreased (Investigations) | 8 | 11
Decreased appetite (Metabolism and nutrition disorders) | 42 | 30
Dehydration (Metabolism and nutrition disorders) | 3 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 8
Dizziness (Nervous system disorders) | 9 | 12
Headache (Nervous system disorders) | 54 | 54
Neuropathy peripheral (Nervous system disorders) | 8 | 4
Paraesthesia (Nervous system disorders) | 6 | 8
Anxiety (Psychiatric disorders) | 4 | 7
Depression (Psychiatric disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 8 | 11
Proteinuria (Renal and urinary disorders) | 21 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 39 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 10 | 9
Hypertension (Vascular disorders) | 60 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study, for review and comment at least 45 days in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).